CLINICAL TRIAL: NCT04481672
Title: Pilot and Feasibility Study of Intravenous Magnesium in Patients Receiving Hyperthermic Intraoperative Chemotherapy With Cisplatin (HIOCC)
Brief Title: Intravenous Magnesium in Patients Receiving Cisplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Shruti Gupta, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-801
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; Magnesium Sulfate; intraoperative cisplatin
MeSH Terms: conditions — Mesothelioma | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Magnesium Sulfate (Experimental): Starting the night before surgery participants will receive intravenous infusion of magnesium over approximately 36 hours. Dosage amounts will vary among participants as the study is determining the highest dose of magnesium that can be administered safely without severe or unmanageable side effects. The first 5 participants of the study will all receive the same dose of magnesium. The decision to test other doses of magnesium in 5 additional participants will depend on magnesium levels and dose tolerance outcomes in the first 5 participants.
  Participants will be followed for 4 days and undergo blood test to measure magnesium levels at the time of hospital admittance, the morning prior to the surgery, twice immediately after surgery, and twice a day for 3 days after the surgery.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Intravenous infusion of magnesium sulfate prior to intraoperative chemotherapy with cisplatin.

SUMMARY:
This research study, is trying to determine the highest dose of magnesium that can be given safely to people with malignant mesothelioma receiving intraoperative chemotherapy with cisplatin who are at risk for acute kidney injury.

The name(s) of the study drug involved in this study is

* magnesium sulfate.

DETAILED DESCRIPTION:
This research study is a phase 1 pilot study, which is the first time investigators are examining larger doses of magnesium in patients receiving cisplatin and the effect of intravenous magnesium administration on blood magnesium levels. In previous studies it was found that patients with lower blood magnesium levels were at higher risk of acute kidney injury. The study is looking to determine the best dose(s) of intravenous magnesium to administer safely without severe or unmanageable side effects in participants. The purpose of the study is also to determine the dose of intravenous magnesium needed to achieve a target level.

The U.S. Food and Drug Administration (FDA) has not approved magnesium for people with mesothelioma receiving cisplatin but it has been approved for other uses.

The research study procedures include: screening for eligibility and study treatment at participant's preoperative visit with their thoracic surgeon. Intravenous magnesium will be administered in the hospital, the night prior to surgery, and take place over 36 hours. Participants will followed for 4 days on postoperative days 1, 2, and 3.

It is expected that about 10 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with malignant mesothelioma admitted for HIOCC. Because no dosing or adverse event data are currently available on the use of intravenous magnesium participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric studies.
* Glomerular filtration rate (GFR)≥ 30 ml/min/1.73m2 at the time of enrollment
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with a pre-treatment serum Magnesium level >2.5 mg/dl or <1.3 mg/dl at the preoperative visit
* Patients with AKI at the time of enrollment, assessed by Kidney Disease Improving Outcomes Criteria (serum creatinine increase ≥1.5x baseline)
* Patients with estimated glomerular filtration rate <30 ml/min/1.73m2 at the time of enrollment
* Patients with neuromuscular disease (e.g., amyotrophic lateral sclerosis, multiple sclerosis, muscular dystrophy, myasthenia gravis, myositis)
* Patients with sustained bradycardia (heart rate <50 beats per minute on 1 or more EKGs in the preceding 90 days) or 2nd degree AV heart block type 2 or higher with the absence of a functioning pacemaker
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to intravenous magnesium
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because they may need magnesium for treatment of preeclampsia or eclampsia, apart from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability as measured by participant rates of enrollment | 6 months
  Feasibility assessed by % of patients that agree to participate. Project feasible if >30% of the patients approached agree to participate
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Time of magnesium infusion till 2 days.
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Magnesium Level | Day of surgery through postoperative day 3.
  Assess the amount of IV magnesium needed to reach a target level of 3 to 4.8mg/dl. Magnesium levels will be measured at multiple time points. We want >80% (≥32/40) of the time-averaged, postoperative magnesium levels to be within the target range of 3 to 4.8 mg/dl.
Tubular Injury Markers | From admission through postoperative day 3
  Changes in urinary KIM-1 and urinary NGAL levels in order to assess intra- and interassay variability

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Gupta, MD, MPH, Principal Investigator — Brigham and Women's Hospital; David E. Leaf, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu